CLINICAL TRIAL: NCT00463281
Title: Observational Study of Multimodal CT in Acute Ischemic Stroke to Define a Tissue Window for Thrombolysis
Brief Title: CT Based Definition of a Tissue Window for Acute Stroke Thrombolysis
Acronym: CT-DEFINE
Status: Completed | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Imanuel Dzialowski, MD, University of Dresden
Other Study IDs: 23211204
Record Dates: First submitted 2007-04-19; First posted 2007-04-20 (Estimated); Last update posted 2009-05-14 (Estimated); Status verified 2009-01

CONDITIONS: Stroke
Keywords: stroke, ischemic; computed tomography; thrombolysis
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Aim of this study is to define a CT-based "tissue window" for stroke thrombolysis. Our primary hypothesis is that

1. patients with a "tissue window" (favourable non-contrast CT (NCCT) scan and an intracranial occlusion on CT angiography (CTA) or perfusion-CT-mismatch" (area of reduced cerebral blood flow (CBF) > area of reduced cerebral blood volume (CBV)) represent a significant proportion (> 20%)of acute stroke patients and therefore are an important target group for future interventional studies
2. patients with a "tissue window" suffer an unfavourable outcome (> 50 % mRS =>4 at 3 months)if the occluded artery was not recanalized.

ELIGIBILITY:
Inclusion Criteria:

* ischemic anterior circulation stroke
* last seen normal < 12 hours
* stroke severity => 3 on the National Institute of Health Stroke Scale
* multimodal CT stroke protocol performed
* informed consent obtained

Exclusion Criteria:

* premorbid modified Rankin Scale score > 3
* contraindications to contrast media application
* pregnancy or breast feeding
* subacute stroke > 50 % of MCA territory
* CT evidence of non-vascular cause of stroke symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ischemic stroke patients presenting within 12 hrs from symptom onset
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2007-01; Primary Completion 2008-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
modified Rankin Scale scores 0-2 | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Imanuel Dzialowski, MD, Principal Investigator — University of Dresden, Dept of Neurology
Locations (1):
- University of Dresden, Dept of Neurology, Dresden, Germany

REFERENCES:
- [Background] Pepper EM, Parsons MW, Bateman GA, Levi CR. CT perfusion source images improve identification of early ischaemic change in hyperacute stroke. J Clin Neurosci. 2006 Feb;13(2):199-205. doi: 10.1016/j.jocn.2005.03.030. Epub 2006 Feb 3. PMID 16459089
- [Background] Parsons MW, Pepper EM, Bateman GA, Wang Y, Levi CR. Identification of the penumbra and infarct core on hyperacute noncontrast and perfusion CT. Neurology. 2007 Mar 6;68(10):730-6. doi: 10.1212/01.wnl.0000256366.86353.ff. PMID 17339580
- [Background] Hill MD, Rowley HA, Adler F, Eliasziw M, Furlan A, Higashida RT, Wechsler LR, Roberts HC, Dillon WP, Fischbein NJ, Firszt CM, Schulz GA, Buchan AM; PROACT-II Investigators. Selection of acute ischemic stroke patients for intra-arterial thrombolysis with pro-urokinase by using ASPECTS. Stroke. 2003 Aug;34(8):1925-31. doi: 10.1161/01.STR.0000082483.37127.D0. Epub 2003 Jul 3. PMID 12843342